CLINICAL TRIAL: NCT05946564
Title: A Multicenter Randomized Trial to Evaluate the Efficacy of Pioglitazone to Promote Renal Tolerance in ANCA-associated Vasculitis - RENATO
Brief Title: A Trial to Evaluate the Efficacy of Pioglitazone to Promote Renal Tolerance in ANCA-associated Vasculitis - RENATO Trial
Acronym: RENATO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP211045; 2022-501057-36-00 (Other: EU CT Number); PHRC-20-0707 (Other Grant/Funding Number: French ministry of health)
Record Dates: First submitted 2023-06-06; First posted 2023-07-14 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: ANCA Associated Vasculitis; Rapidly Progressive Glomerulonephritis; Crescentic Glomerulonephritis
Keywords: ANCA; vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis | interventions — Pioglitazone

STUDY DESIGN:
Intervention Model Description: Comparative, multicentre, prospective, randomized, placebo-controlled double-blind phase III trial, evaluating the efficacy of add-on pioglitazone therapy on top of a standard of care (SOC) immunosuppressive therapy, in patients with ANCA-associated vasculitis and biopsy-proven renal involvement. Patients eligible for the study will be assigned in a 1:1 randomized fashion to additional treatment by pioglitazone (30 mg/day orally) or to placebo for 26 weeks on top of a SOC immunosuppressive treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind (investigators and patients)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pioglitazone (ACTOS®) (Experimental): Pioglitazone given once a day, orally, at 30 mg dose, for 26 weeks
  Interventions: Drug: Pioglitazone (ACTOS®)
- Placebo of pioglitazone (Placebo Comparator): Placebo of pioglitazone, given once a day, orally, for 26 weeks
  Interventions: Drug: Placebo of Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone (ACTOS®) — Patient will be randomize in the intervention group receive treatment by pioglitazone (30 mg/day orally) for 26 weeks on top of a SOC immunosuppressive treatment.
  Arms: Pioglitazone (ACTOS®)
Drug: Placebo of Pioglitazone — Patient will be randomize in the intervention group receive treatment by placebo of pioglitazone (30 mg/day orally) for 26 weeks on top of a SOC immunosuppressive treatment.
  Arms: Placebo of pioglitazone

SUMMARY:
The RENATO trial is a multicenter randomized controlled trial that evaluates the efficacy of pioglitazone to improve renal outcomes in ANCA-associated vasculitis.

Patients with biopsy-proven kidney involvement of ANCA vasculitis will be included in this trial at diagnosis. All patients will receive a standard of care immunosuppressive (SOC) therapy combining corticosteroids and rituximab (375 mg/m2/week for 4 consecutive weals followed by 500 mg re-infusion every 6 months). They will be randomized 1:1 to receive either pioglitazone 30 mg/day or placebo for 6 months, on top of SOC. The primary objective of this trial is to demonstrate that pioglitazone reduces kidney damage, reflected by the early improvement of proteinuria and serum creatinine levels. The secondary objectives will be to assess the efficacy of this drug on the reduction of hypertension and metabolic effects of glucocorticoids, to measure its impact on vasculitis activity and to evaluate the safety profile of pioglitazone in this population.

DETAILED DESCRIPTION:
After a patient has consented to participate to the study, the informed consent form will be signed by the patient and the investigator. The patient will be randomized to one of two groups (pioglitazone or placebo). The patient will take the experimental treatment for 26 weeks and his research follow-up will last 52 weeks (follow-up visit : W1, W2, W3, W4 (research visit), W8, W12, W26, W38 and W52).

All participants will receive SOC immunosuppressive treatment with rituximab at 375 mg/m2/week for 4 consecutive weeks, as induction therapy of vasculitis flare, followed by 500 mg re-infusion every 6 months/24 weeks as maintenance therapy, i.e. at week 26 and 52, as recommended. The two treatment groups will also receive a standardized glucocorticoid tapering schedule: one to three i.v. pulses of methylprednisolone (7.5 to 15 mg/kg each) according to physician decision, followed by a predefined oral prednisone tapering schedule as used in the reduced-dose arm of the PEXIVAS trial.

Samples (plasma, serum and urine) taken as part of the study will be stored in a biological sample collection (at D0, W1, W2, W3, W12, W26, W38 and W52 visits).

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed or relapsing ANCA-associated vasculitis, i.e. granulomatosis with polyangitis (GPA) or microscopic polyangiitis (MPA), according to ACR 1990 criteria and/or revised Chapel Hill Consensus Conference definitions and/or European Medical Agency algorithm, with an active disease defined as a BVAS ≥3
* Presence of proteinuria (UPCR >300 mg/g), haematuria (>10 RBC/hpf), and eGFR ≥15 mL/min/1.73 m2 (CKD-EPI formula) at inclusion (<1 month)
* Recent (<4 weeks) renal biopsy that confirms active renal involvement of ANCA-associated vasculitis
* Patients aged of 18 to 80 years
* Participant written informed consent prior to participation in the study
* Participants affiliated to a French health insurance system (registered or being a beneficiary of such a scheme)

Exclusion Criteria:

* Alveolar haemorrhage requiring pulmonary ventilation support at inclusion
* Patients with eosinophilic granulomatosis with polyangiitis (EGPA, Churg-Strauss)
* Active cancer (except non-melanoma skin cancer) within the past 24 months
* Active severe bacterial, viral or fungal infectious disease
* Past history of bladder or urinary tract cancer
* History of Class 3/4 congestive heart failure symptoms, any time
* History of Class 2 heart failure symptoms within the past 3 months and/or ejection fraction <40% on recent echocardiography (<1 month)
* Transaminases levels above 2 times the normal range value (<1 month) or any severe chronic liver disease
* Positive serology for HIV, HBV (Ag HBs positivity) or active HCV infection at inclusion
* Presence of neutropenia <1000 cells/l (<1 month)
* History of intolerance to any thiazolidinedione (including Pioglitazone), to rituximab or any excipient listed in SmPc
* Diabetic ketoacidosis, any time
* A pre-existing or an important risk of new-onset macular edema (confirmed by an ophthalmological examination)
* Pregnant or breast-feeding women, or desire to become pregnant within 24 months All women of childbearing potential (WOCBP) are required to have a negative pregnancy test before treatment and must agree to maintain highly effective contraception by practicing abstinence or by using an effective method of birth control from the date of consent through the end of the study and another 12 months after (or 12 months after the last rituximab infusion in case of premature termination): Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (Oral, Intravaginal, Transdermal); Progestogen-only hormonal contraception associated with inhibition of ovulation (Oral, Injectable, Implantable); Intrauterine device (IUD); Intrauterine hormone-releasing system (IUS); Bilateral tubal occlusion; Vasectomised partner
* Severe neurologic or psychiatric disease (e.g., dementia or schizophrenia)
* Kidney transplant recipients
* Cyclophosphamide or rituximab (dose > 375 mg/m2) use within 26 weeks prior to screening; if on azathioprine, mycophenolate mofetil or methotrexate at the time of screening, these drugs must be withdrawn prior to receiving the first rituximab dose. Patients that have initiated induction therapy with rituximab for the actual flare, can be included in the present study within 48h following the first rituximab infusion
* Intravenous glucocorticoids, >3000 mg methylprednisolone equivalent, within 4 weeks prior to screening
* Patients who have been taking an oral daily dose of a glucocorticoid of more than 10 mg prednisone-equivalent for more than 6 weeks continuously prior to screening
* Current participation in another research study involving a therapeutic intervention. Participation to an observational research, or a non-interventional research is allowed
* Patients under guardianship or curators and protected adults
* Patients not able to understand and follow study procedures
* Patients on AME (Aide Médicale de l'Etat = State Medical Assistance)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2027-04-24 (Estimated); Study Completion 2027-10-24 (Estimated)

PRIMARY OUTCOMES:
Appearance of a success defined as (1) Delta sCreat > 30% (between D0 and week 26) AND (2) urine protein-to-creatinine (uPCR) < 1g/mmol | Week 26

SECONDARY OUTCOMES:
Change of renal function | Weeks 4, 12, 26 and 52
  Delta sCreat (baseline sCreat - follow-up sCreat)
Proteinuria ratio | Weeks 4, 12, 26 and 52
  Spot urine protein-to-creatinine ratio (uPCR)
Score VDI (Vasculitis Damage Index) | Week 26 and 52
  Systemic chronic damage due to vasculitis and treatment of vasculitis Min : 0 Max : 62 the best score is 0
Renal vasculitis activity | Weeks 4, 12, 26 and 52
  measurement of urine biomarkers: MCP-1
Renal vasculitis activity | Weeks 4, 12, 26 and 52
  measurement of urine biomarkers: KIM-1
Renal vasculitis activity | Weeks 4, 12, 26 and 52
  measurement of urine biomarkers: Calprotectin
Renal vasculitis activity | Weeks 4, 12, 26 and 52
  measurement of urine biomarkers: CD163
Systemic vasculitis activity : score BVAS | Weeks 4, 12, 26 and 52
  BVAS (Birmingham Vasculitis Activity Score ), ANCA positivity Min : 0 Max : 63 The best score is 0
Refractory vasculitis | Weeks 12, 26 and 52
  Percentage of patients with refractory vasculitis and early vasculitis relapses
Improvement in Quality of Life (SF-36) | baseline, weeks 4, 12, 26 and 52
  SF-36 : Short-form 36 Min : 0 Max : 100 A low score reflects a perception of poor health, loss of function, presence of pain. A high score reflects a perception of good health, an absence of functional deficit and pain.
Improvement in Quality of Life (EQ-5D) | baseline, weeks 4, 12, 26 and 52
  EQ-5D : Euroqol Min: 0 Max : 100 Higher scores mean a better
Safety profile of pioglitazone | Weeks 26 and 52
  numbers of adverse events, numbers of patients with adverse events, numbers of serious adverse events
Toxicity induced by glucocorticoids | Weeks 12, 26 and 52
  Glucocorticoid Toxicity Index (GTI) the best score is 0
Change metabolic effects of Glucocorticoids | Weeks 12, 26 and 52.
  To assess the efficacy of pioglitazone on the reduction metabolic side effects of glucocorticoids by HbA1c
Change metabolic effects of Glucocorticoids | Weeks 12, 26 and 52.
  To assess the efficacy of pioglitazone on the reduction metabolic side effects of glucocorticoids by evaluation of lipid profile
Change blood pressure | Weeks 12 and 26.
  To assess the efficacy of pioglitazone on the reduction of hypertension)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Karras, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (24):
- France (24):
  - CHU Amiens, Amiens
  - CHU d'Angers, Angers
  - CH de Boulogne sur Mer, Boulogne-sur-Mer
  - CHU Brest - Hôpital de la Cavale Blanche, Brest
  - CHU de Dijon, Dijon
  - CHU de Grenoble - Hôpital Michalon site nord, Grenoble
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Hopital Le Kremlin Bicetre - Aphp, Le Kremlin-Bicêtre
  - AP-HM - Hôpital la Conception, Marseille
  - CHU de Nantes - Hotel Dieu, Nantes
  - CHU Pasteur 2 - Nice, Nice
  - CHU Nîmes - Hôpital universitaire Caremeau, Nîmes
  - AP-HP - Hôpital Cochin, Paris
  - AP-HP - Necker enfants malades, Paris
  - HEGP, Paris
  - AP-HP - Hôpital Bichat, Paris
  - AP-HP - Tenon, Paris
  - AP-HP - Henri Mondor, Paris
  - CHU de Rouen, Rouen
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse - Hôpital Rangueil, Toulouse
  - CH Valenciennes, Valenciennes
  - Chru de Nancy, Vandœuvre-lès-Nancy
  - Hôpital Robert Schuman (UNEOS), Vantoux

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).